CLINICAL TRIAL: NCT03196947
Title: Phase I, Open Label, Dose Escalation Study to Investigate the Tolerability and Efficacy of APO010 in Patients With Relapsed/Refractory Multiple Myeloma Selected by Drug Response Predictor (DRP)
Brief Title: Safety and Pharmacokinetics of Rising Doses of APO010 in Relapsed/Refractory Multiple Myeloma Patients Selected by DRP
Acronym: SMR-3184
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to sponsors decision
Sponsor: Allarity Therapeutics (Industry)
Collaborators: Smerud Medical Research International AS (Other); Medical Prognosis Institute A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APO010/P1/002
Record Dates: First submitted 2017-05-19; First posted 2017-06-23 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: multiple myeloma; APO010; Drug Response Predictor; DRP
MeSH Terms: conditions — Multiple Myeloma | interventions — Mega-Fas-ligand

STUDY DESIGN:
Intervention Model Description: Dose Escalation followed by an extension phase using the recommended dosage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm, APO010 Dose escalation (Experimental)
  Interventions: Drug: APO010

INTERVENTIONS:
Drug: APO010 — APO010 is given iv on D1, D8 and D15 followed by a one-week drug rest (cycle duration 4 weeks).

SUMMARY:
Multicentre, open label, uncontrolled, phase I pharmacokinetic study, to determine the Maximum Tolerated Dose (MTD) of APO010 administered intravenously on D1, D8 and D15 followed by a one-week drug rest, in patients with multiple myeloma for who have relapsed or are refractory to 2 (in high-risk patients 1) or more different prior therapies and who have Drug Response Predictor (DRP) for APO010 indicating a higher likelihood for response to APO010. The study will contain an extension phase where the recommended Dose will be tested on additional patients.

DETAILED DESCRIPTION:
APO010 is a novel investigational antitumour agent. It is a recombinant form of human Fas ligand (FasL), a protein with the function of inducing programmed cell death (apoptosis). Preclinical studies indicate that multiple myeloma is sensitive for APO010. Estimation of DRP for APO010 in myeloma patients suggests that it may be possible to identify patients with high and low likelihood for response, and thereby allocate the predicted high likelihood patients to the treatment. Preclinical results indicate that, in comparison with other single agents, APO010 exercises superior anti-tumour effect by inducing apoptosis.

The study will include patients with multiple myeloma who have relapsed or are refractory to 2 (in high-risk patients 1) or more different prior therapies, including IMiDs and PI and who have Drug Response Predictor (DRP) for APO010 indicating a higher likelihood for response to APO010.

This study is a multicentre, open label, uncontrolled, phase I, dose escalation, pharmacokinetic study, to determine the Maximum Tolerated Dose (MTD) of APO010 administered intravenously on D1, D8 and D15 followed by a one-week drug rest i.e. cycle duration is 4 weeks. The study will contain an extension phase where the Recommended Dose will be tested on additional patients.

The primary endpoint is determination of the Maximum Tolerated Dose (MTD)based upon first cycle drug-related dose-limiting toxicity and the recommended dose of APO010. Safety will be evaluated during the study and for 30 days after the last administration of study drug. Adverse events and laboratory studies will be graded according to NCI-CTCAE v. 4.03.

The proportion of patients with positive HADA assessment will be investigated and a description of any objective tumour response based on International Myeloma Working Group criteria and from changes in M-protein and iFLC.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or relapsed/refractory to 2 (in high-risk patients 1) or more different prior therapies, including IMiDs and PI
* Measurable disease
* Serum M-protein > 10 g/l, or
* Urine M-protein > 200 mg/24 hours, or
* Serum involved-FLC (iFLC) > 100 mg/l and abnormal FLC ratio
* Have participated in the APO010 screening protocol in which Drug Response Predictor (DRP) outcome is measured as being in the upper likelihood of response (50% in dose-finding part and 25% in the expansion cohort)
* Age > 18 years
* Adequate organ and bone marrow function as defined below:
* Absolute neutrophil count > 1.5 x 109/l (> 0.75 x 109/l in case > 50% plasma cell count in bone marrow)
* Platelet count > 50 x 109/l (> 30 x 109/l in case > 50% plasma cell count in bone marrow)
* Haemoglobin > 4.6 mmol/l (> 7.5 g/l)
* Bilirubin ≤ upper limit of normal
* aspartate aminotransferase (SGOT)/alanine transaminase (SGPT) ≤ upper limit of normal
* Creatinine < 1.5 x upper limit of normal or creatinine clearance > 50 ml/min calculated according to Cockcroft-Gault
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Life expectancy of at least 3 months.
* Capability of understanding the nature of the study and giving written informed consent
* Signed informed consent form

Exclusion Criteria:

* Have central nervous system (CNS) myeloma
* Have plasma cell leukaemia defined as plasma cell count > 2000 / µL in peripheral blood
* Have symptomatic amyloidosis
* Have anti-myeloma treatment or radiotherapy within 3 weeks from first infusion
* Have received a cumulative dose of corticosteroid > 200 mg (dexamethasone, or equivalent dose of prednisone) within 2 weeks of the first infusion
* Have received any experimental drug or experimental therapy within 3 weeks before the first infusion
* Have received autologous-stem cell transplantation (SCT) within 12 weeks before the first infusion
* Have received an allogeneic stem cell transplantation (SCT)
* Have had past or current malignancy except for:
* Cervical carcinoma < Stage 1B
* Non-invasive basal cell or squamous cell skin carcinoma
* Malignant melanoma with CR of > 10 years
* Any other curable cancer with a CR > 5 years
* Have major surgery within 4 weeks prior to the first infusion
* Have severe infection requiring iv treatment
* Have known HIV positivity
* Have known active hepatitis B or C
* Have had clinical significant arteriosclerotic events:
* Ischemic heart disease
* Unstable angina
* Myocardial infarction
* Transient ischemic attack
* Ischemic stroke
* Documented peripheral arteriosclerosis
* Have baseline QT interval as corrected by Fridericia's formula (QTcF) > 470 msec for female patients or > 450 msec for male patients or a complete left bundle branch block (defined as QRS interval > 120 msec in left bundle branch block form)
* CNS disease including epilepsy or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures
* Women of childbearing age and potential who are not willing to use effective contraception during the study and at least until 90 days after last dose of study drug. Male patients or male patients who have female partners of childbearing age and potential who are not willing to use effective contraception during the study and at least until 90 days after last dose of study drug. Highly effective methods of birth control are defined as those which result in a low failure rate, i.e., less than 1% per year, when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra-uterine devices, sexual abstinence or vasectomized partner
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dosage | 1 Year
  To define the Maximum Tolerated Dosage of intravenous bolus administration of APO010
Recommended Dosage | 1 Year
  To define the Recommended Dosage of intravenous bolus administration of APO010

SECONDARY OUTCOMES:
Percentage (%) of patients with drug-related adverse events (adverse reactions) | 1 Year
  To define the safety profile of a weekly schedule of APO010, including Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.03, Physical examination, vital signs, concomitant medications and laboratory data. To define the safety profile of APO010 after chronic administration (beyond 3 consecutive administrations, i.e., two or more cycles) and to define local toxicity at the site of administration through observation of the area of infusion.
The pharmacokinetic profile (AUC INF) for APO010 at doses above 60 µg/m2 | 1 Year
  The PK variable that will be evaluated are Area Under the curve (AUC INF). Pharmacokinetic parameters will be measured for APO010 at doses above 60 µg/m2
The pharmacokinetic profile (AUC last) for APO010 at doses above 60 µg/m2 | 1 Year
  The PK variable that will be evaluated are Area Under the curve (AUC last). Pharmacokinetic parameters will be measured for APO010 at doses above 60 µg/m2
The pharmacokinetic profile (AUC 0-12hr) for APO010 at doses above 60 µg/m2 | 1 Year
  The PK variable that will be evaluated are Area Under the curve (AUC 0-12hr). Pharmacokinetic parameters will be measured for APO010 at doses above 60 µg/m2
The Maximum Plasma Concentration (Cmax), for APO010 at doses above 60 µg/m2 | 1 Year
  The PK variable that will be evaluated is Maximum Plasma Concentration (Cmax). Pharmacokinetic parameters will be measured for APO010 at doses above 60 µg/m2
The Observed maximum (Tmax), for APO010 at doses above 60 µg/m2 | 1 Year
  The PK variable that will be evaluated is, time of observed maximum (Tmax). Pharmacokinetic parameters will be measured for APO010 at doses above 60 µg/m2
The Terminal half-life (T½), for APO010 at doses above 60 µg/m2 | 1 Year
  Pharmacokinetic (PK) parameters will be calculated or estimated by using a model independent approach. The PK variable that will be evaluated is the terminal half-life (T½)). Pharmacokinetic parameters will be measured for APO010 at doses above 60 µg/m2
The HADA Antibody Response | 1 Year
  Assays will be performed to detect the production of antibodies against APO010 (HADA) in the serum of treated patients. If antibodies are formed, their ability to neutralize the biological activity of APO010 in in vitro cytotoxicity assay will be measured.
The Tumor Response | 1 Year
  Using International Myeloma Working Group (IMWG) response criteria, based on measurements in blood and urine and in case of disappearance of M-proteins with additional confirmatory bone-marrow investigation, the number of patients with either stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), stable disease (SD) or progressive disease (PD) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Annette J Vangsted, DMSc, Principal Investigator — Rigshospitalet, Finsen Centre, Hematological Department,, Phase 1 Unit
Locations (1):
- University Hospital of Copenhagen, Copenhagen, Denmark